CLINICAL TRIAL: NCT06514638
Title: Computational Mathematical Analysis of the Texture of Muscle Tissue in Vastus Medialis Between a MTrP and a Non-painful Point
Brief Title: Computational Mathematical Analysis in Vastus Medialis Between a MTrP and Non Painful Point
Status: Completed | Type: Observational
Sponsor: Samuel Fernández Carnero (Other)
Responsible Party: Sponsor-Investigator, Samuel Fernández Carnero, Physical Therapy PhD, University of Alcala
Organization: University of Alcala (Other)
Other Study IDs: Vastus ultrasound MTRp
Record Dates: First submitted 2024-07-11; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: ultrasound; myofascial trigger point; vastus medialis
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study subjects: Helathy, 18-65 year old subjects with pain when fingerr pointed in the vastus medialis, without serious diseases.
  Interventions: Other: Ultrasound imaging

INTERVENTIONS:
Other: Ultrasound imaging — Images of the vastus medialis were taken with the subject being lateral decubitus.

SUMMARY:
With the help of ultrasound, the goal of the study is to asses the differences between MTR points and non painful points, in order to characterize the identification of MTR througought ultrasound. Being a complex process that needs to be standarized for each muscle, the study takes place in the vastus medialis.

DETAILED DESCRIPTION:
Nowadays, myofascial trigger points (MTrP) represent one of the most common musculoskeletal alterations in clinic, being many times diffuse and complex to diagnose and localize. Ultrasound is a therapeutic tool used in physiotherapy for assessment and treatment. Some of its advantages include the quickness and harmlessness. Linking these two concepts, there is no vast evidence regarding the identification of myofascial trigger points through ultrasound. A computational mathematical analysis was performed throughout ultrasound images of the vastus medialis in order to characterize MTrPs, where images of 66 participants vastus medialis were taken. Two investigators made the finger point palpation locating a MTrP and a non-painful point. A third investigator screened the photographs with the ultrasound and a preset for the zone. 3 images were taken from the MTrP, 3 from the non-painful point, and other 3 of a different MTrP, in case the investigators disagreement of the MTrP location. A fourth investigator carried out the histogram analysis using Fiji software. Lastly, stastistical analysis of the study variables was performed.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 year old.
* Presence of pain on palpation along the course of the muscle fibers of the vastus medialis of the quadriceps.
* Painful point and/or localized tense band with or without radiation of pain to the knee area or adductor region.

Exclusion Criteria:

* Serious diseases (neurological, psychiatric, systemic diseases, obesity).
* Knee or hip surgeries.
* Muscle tears in a state of recovery in the vastus medialis of the quadriceps.
* Inability to position yourself in a lateral decubitus position.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Students in the university were the main collection of subjects because of the proximity, but also other people recruited around the city.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-06-23 (Actual)

PRIMARY OUTCOMES:
Echogenicity | Through study completion, an average of 3 months
  Information measures of correlation at 0º, 45º, 90º, 135º expressed as mean+-standard deviation

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Tercero Mendoza, BSc, Principal Investigator — University of Alcala; David Hernández Sánchez, BSc, Principal Investigator — University of Alcala; Daniel Roldán Peña, BSc, Principal Investigator — University of Alcala; Noe López Castellanos, BSc, Principal Investigator — University of Alcala
Locations (1):
- Nursing and Physiotherapy Faculty Study Officials, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Yet to be decided, maybe collected as a part of a protocol to standarize.

REFERENCES:
- [Background] Sikdar S, Shah JP, Gebreab T, Yen RH, Gilliams E, Danoff J, Gerber LH. Novel applications of ultrasound technology to visualize and characterize myofascial trigger points and surrounding soft tissue. Arch Phys Med Rehabil. 2009 Nov;90(11):1829-38. doi: 10.1016/j.apmr.2009.04.015. PMID 19887205
- [Background] Hsieh CY, Hong CZ, Adams AH, Platt KJ, Danielson CD, Hoehler FK, Tobis JS. Interexaminer reliability of the palpation of trigger points in the trunk and lower limb muscles. Arch Phys Med Rehabil. 2000 Mar;81(3):258-64. doi: 10.1016/s0003-9993(00)90068-6. PMID 10724067
- [Background] Rathbone ATL, Grosman-Rimon L, Kumbhare DA. Interrater Agreement of Manual Palpation for Identification of Myofascial Trigger Points: A Systematic Review and Meta-Analysis. Clin J Pain. 2017 Aug;33(8):715-729. doi: 10.1097/AJP.0000000000000459. PMID 28098584
- [Background] Martinez-Paya JJ, Rios-Diaz J, Del Bano-Aledo ME, Tembl-Ferrairo JI, Vazquez-Costa JF, Medina-Mirapeix F. Quantitative Muscle Ultrasonography Using Textural Analysis in Amyotrophic Lateral Sclerosis. Ultrason Imaging. 2017 Nov;39(6):357-368. doi: 10.1177/0161734617711370. Epub 2017 May 28. PMID 28553752
- [Background] Kumbhare DA, Elzibak AH, Noseworthy MD. Assessment of Myofascial Trigger Points Using Ultrasound. Am J Phys Med Rehabil. 2016 Jan;95(1):72-80. doi: 10.1097/PHM.0000000000000376. PMID 26334421
- [Background] Nadeau MJ, Desrochers A, Lamontagne M, Lariviere C, Gagnon DH. Quantitative ultrasound imaging of Achilles tendon integrity in symptomatic and asymptomatic individuals: reliability and minimal detectable change. J Foot Ankle Res. 2016 Aug 17;9:30. doi: 10.1186/s13047-016-0164-3. eCollection 2016. PMID 27540416
- [Background] Stock MS, Thompson BJ. Echo intensity as an indicator of skeletal muscle quality: applications, methodology, and future directions. Eur J Appl Physiol. 2021 Feb;121(2):369-380. doi: 10.1007/s00421-020-04556-6. Epub 2020 Nov 21. PMID 33221942
- [Background] Schindelin J, Arganda-Carreras I, Frise E, Kaynig V, Longair M, Pietzsch T, Preibisch S, Rueden C, Saalfeld S, Schmid B, Tinevez JY, White DJ, Hartenstein V, Eliceiri K, Tomancak P, Cardona A. Fiji: an open-source platform for biological-image analysis. Nat Methods. 2012 Jun 28;9(7):676-82. doi: 10.1038/nmeth.2019. PMID 22743772
- See also: 1. Borg-Stein, J., & Iaccarino, M. A. (2014). Myofascial pain syndrome treatments. Physical medicine and rehabilitation clinics of North America — https://doi.org/10.1016/j.pmr.2014.01.012